CLINICAL TRIAL: NCT07297719
Title: A Non-interventional, Single-visit Study Focusing on the Evaluation of Glistening as Well as General Safety and Visual Outcomes With at Least 24 Months Follow-up in Patients Implanted With CT LUCIA 621P Intraocular Lenses
Brief Title: Evaluation of Glistening, Visual Outcomes and General Safety 24 Months Post-IOL Implantation
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CT LUCIA 621P-BER-401-25
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Cataract Senile
Keywords: IOL; Glistening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Main evaluation of glistening at least 24 Months post-IOL implantation

DETAILED DESCRIPTION:
Evaluation of glistening, visual outcomes and general safety after at least 24 Months post-IOL implantation

ELIGIBILITY:
Inclusion Criteria:

1. Patients currently implanted with the CT LUCIA 621P IOL into the capsular bag in at least one eye and who participated in previous study "CT LUCIA 621P-BER-401-21";
2. A minimum follow-up period of 24 months after the IOL implantation of the study eye (selected as the study eye in the previous study);
3. Patients willing and capable of providing informed consent;
4. Patients willing and capable of complying with visits and procedures as defined by this protocol.

Exclusion Criteria:

1. Complications during cataract surgery with clinically significant impact;
2. Postoperative clinically significant corneal or retinal pathology as well as postoperative acute or chronic inflammatory ocular conditions (e.g. uveitis, iritis etc.);
3. Presence of clinically significant PCO with potential to limit the glistening evaluation;
4. IOL dislocation (the complete IOL is not stable fixated in the capsular bag);
5. Patients unable to meet the limitations of the protocol or likely of non-cooperation during the clinical investigation;
6. Patients whose freedom is impaired by administrative or legal order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently implanted with the CT LUCIA 621P IOL from the Aier Eye Hospital of BoAo Hope City
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2025-12-25 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Glistening Evaluation | 24 months post IOL Implantation
Monocular Corrected Distance Visual Acuity (CDVA) | 24 months post IOL Implantation
  Evaluation of the monocular Corrected Distance Visual Acuity (CDVA) a

OTHER OUTCOMES:
Monocular uncorrected distance visual acuity (UDVA) | 24 months post IOL Implantation
Refraction | 24 months post IOL Implantation
Refraction predictability | 24 months post IOL Implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Aier Eye Hospital of BoAo Hope City, Hainan, Hainan, China

IPD SHARING:
Plan to Share IPD: No